CLINICAL TRIAL: NCT05934630
Title: CSF Cell-free Tumor DNA (CSF cfDNA) Liquid Biopsies for Pediatric, Adolescent, and Young Adult Patients With Primary Brain Tumors
Brief Title: Testing Cerebrospinal Fluid for Cell-free Tumor DNA in Children, Adolescents, and Young Adults With Brain Tumors
Status: Suspended | Type: Observational
Why Stopped: Memorial Sloan Kettering Cancer Center (MSKCC) is undergoing institutional system updates and has requested the hold.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Other Study IDs: PBTC-N14; UM1CA081457 (NIH); NCI-2023-02321 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-N14 (Other: Pediatric Brain Tumor Consortium); PBTC-N14 (Other: CTEP)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Anaplastic Astrocytoma; Diffuse Brainstem Glioma; Glioblastoma Multiforme; High-grade Astrocytoma NOS; Fibrillary Astrocytoma; Low-Grade Astrocytoma, Nos; Pilocytic Astrocytoma; Choroid Plexus Carcinoma; CNS Primary Tumor, Nos; Atypical Teratoid/Rhabdoid Tumor; Medulloblastoma; Supratentorial Primitive Neuroectodermal Tumor; Ependymoma, NOS; Anaplastic Oligodendroglioma; Oligodendroglioma, Nos; CNS Germ Cell Tumor; Pineoblastoma; Diffuse Leptomeningeal Glioneuronal Tumor
Keywords: Liquid biopsy; CSF; Cerebrospinal fluid; cfDNA; ctDNA; Pediatric central nervous system tumors; Brain tumor
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Choroid Plexus Carcinoma; Central Nervous System Neoplasms; Rhabdoid Tumor; Medulloblastoma; Ependymoma; Oligodendroglioma; Pinealoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Stratum 1: Medulloblastoma: Participants in Arm 1 must have diagnosis of Medulloblastoma. All children and adolescent/young adult (AYA) patients <= 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults.
- Stratum 2: High-grade Glioma (IDH-wildtype) or Diffuse Intrinsic Pontine Glioma: Participants in Arm 2 must have diagnosis of High-grade Glioma (IDH-wildtype) or Diffuse Intrinsic Pontine Glioma (DIPG). All children and adolescent/young adult (AYA) patients <= 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults. DIPG patients must meet clinical and imaging requirements for DIPG diagnosis. Patients with newly diagnosed DIPGs, defined as tumors with a pontine epicenter and diffuse involvement of 2/5 or more of the pons, are eligible without histologic confirmation. Patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible for Stratum 2 if the tumors have been biopsied and are proven to be an anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic mixed glioma or fibrillary astrocytoma.
- Stratum 3: Low-grade Glioma IDH-wildtype with multifocal/disseminated and/or leptomeningeal disease: Participants in Arm 3 must have diagnosis of Low-grade Glioma (IDH-wildtype) with multifocal/disseminated and/or leptomeningeal disease. All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults.
- Stratum 4: Diffuse Leptomeningeal Glioneuronal Tumor: Participants in Arm 4 must have diagnosis of Diffuse Leptomeningeal Glioneuronal Tumor. All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults.
- Stratum 5: Pineoblastoma: Participants in Arm 5 must have diagnosis of Pineoblastoma. All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults.
- Stratum 6: All other eligible primary brain tumor types: Participants in Arm 6 must have diagnosis of all other eligible primary brain tumor types. All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults.

SUMMARY:
Recent advances in technology have allowed for the detection of cell-free DNA (cfDNA). cfDNA is tumor DNA that can be found in the fluid that surrounds the brain and spinal cord (called cerebrospinal fluid or CSF) and in the blood of patients with brain tumors. The detection of cfDNA in blood and CSF is known as a "liquid biopsy" and is non-invasive, meaning it does not require a surgery or biopsy of tumor tissue. Multiple studies in other cancer types have shown that cfDNA can be used for diagnosis, to monitor disease response to treatment, and to understand the genetic changes that occur in brain tumors over time. Study doctors hope that by studying these tests in pediatric brain tumor patients, they will be able to use liquid biopsy in place of tests that have more risks for patients, like surgery.

There is no treatment provided on this study. Patients who have CSF samples taken as part of regular care will be asked to provide extra samples for this study. The study doctor will collect a minimum of one extra tube of CSF (about 1 teaspoon or 5 mL) for this study. If the patients doctor thinks it is safe, up to 2 tubes of CSF (about 4 teaspoons or up to 20 mL) may be collected. CSF will be collected through the indwelling catheter device or through a needle inserted into the lower part of the patient's spine (known as a spinal tap or lumbar puncture).

A required blood sample (about ½ a teaspoon or 2 3 mL) will be collected once at the start of the study. This sample will be used to help determine changes found in the CSF. Blood will be collected from the patient's central line or arm as a part of regular care.

An optional tumor tissue if obtained within 8 weeks of CSF collection will be collected if available. Similarities between changes in the DNA of the tissue that has caused the tumor to form and grow with the cfDNA from CSF will be compared. This will help understand if CSF can be used instead of tumor tissue for diagnosis. Up to 300 people will take part in this study.

This study will use genetic tests that may identify changes in the genes in the CSF. The report of the somatic mutations (the mutations that are found in the tumor only) will become part of the medical record. The results of the cfDNA sequencing will be shared with the patient. The study doctor will discuss what the results mean for the patient and patient's diagnosis and treatment. Looking for inheritable mutations in normal cells (blood) is not the purpose of this study. Genetic tests of normal blood can reveal information about the patient and also about the their relatives. The doctor will discuss what the tests results may mean for the patient and the their family. Patient may be monitored on this study for up to 5 years.

DETAILED DESCRIPTION:
This is a multicenter study for children and young adults with primary brain tumor. All children and adolescent/young adult (AYA) patients 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults. Up to 300 people will take part in this study.

Pediatric central nervous system (CNS) tumors represent a wide range of disorders and continue to be the leading cause of cancer-related death in children and adolescents. The past few years have led to a dramatic shift in the diagnosis and pathological classification of pediatric CNS tumors. Molecular biomarkers which are now being incorporated into treatment decisions and clinical trial design. With this, the need for longitudinal molecular monitoring of disease becomes increasingly evident. The anatomical challenges in accessing pediatric CNS malignancies coupled with the move toward molecular sub-classification and molecular targeted therapies leads to an urgent need to develop a non-invasive way to repeatedly sample these tumors. This would enable: 1) diagnose tumors that are surgically inaccessible; 2) monitor molecular changes in tumor longitudinally, including at progression and/or recurrence; and 3) develop non-invasive ways to monitor treatment responses. Recent advances in technology have allowed for the detection of cell-free tumor DNA (cfDNA), i.e., small fragments of tumor DNA, shed into the cerebrospinal fluid (CSF) and bloodstream in brain tumor patients through a process known as "liquid biopsy".

Based on the successful preliminary studies in adult glioma patients, this Pediatric Brain Tumor Consortium (PBTC)-sponsored effort will attempt to integrate CSF cfDNA liquid biopsies into the clinical care of pediatric brain tumor patients across the PBTC to enhance tumor diagnosis/molecular subclassification and guide therapeutic decision making. This will be accomplished through centralized collection and processing of CSF cfDNA samples from patients with various types of pediatric CNS tumors across PBTC member sites. The primary objective will be to investigate the concordance between CSF cfDNA alterations and tumor DNA alterations in matched pairs to understand: 1) the concordance across matched samples; and 2) the genomic evolution that occurs over time across various tumor types. Additionally, the secondary objectives and exploratory objectives in this study are intended to aggregate data across various types of pediatric primary brain tumors to understand the rate of success of CSF cfDNA molecular profiling in different disease types and at various stages of disease, and to elucidate the role of CSF cfDNA profiling in guiding clinical decision making.

The primary objective of this study is to estimate the concordance of mutations detected in the tumor tissue vs. cerebrospinal fluid cell free DNA (CSF cfDNA) across samples collected within 8 weeks of each other; determine whether clonal mutations are likely to be shared across sample types.

Patients who have CSF samples taken as part of regular care will be asked to provide extra samples for this study. The study doctor will collect a minimum of one extra tube of CSF (about 1 teaspoon or 5 mL) for this study. If the patient's doctor thinks it is safe, up to 2 tubes of CSF (about 4 teaspoons or up to 20 mL) may be collected. A required blood sample (about ½ a teaspoon or 2 - 3 mL) will be collected once at the start of the study. An optional tumor tissue if obtained within 8 weeks of CSF collection will be collected if available. There is no treatment provided on this study.

ELIGIBILITY:
Inclusion Criteria:

All patients must have a known or suspected diagnosis (based on pathology or imaging) of a primary brain tumor. All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible.

AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults. This includes:

* medulloblastoma
* non-medulloblastoma embryonal brain tumors
* atypical teratoid rhabdoid tumors (ATRT)
* ependymoma
* CNS germ cell tumors
* Diffuse midline glioma, H3K27M-altered
* Diffuse hemispheric glioma, H3 G34-mutant
* pineoblastoma
* diffuse leptomeningeal glioneuronal tumor
* diffuse brainstem glioma
* pilocytic astrocytoma
* choroid plexus carcinoma

ELIGIBLE PATIENTS WILL BE STRATIFIED BY DIAGNOSIS AS FOLLOWS:

* Stratum 1: Medulloblastoma
* Stratum 2: High-grade glioma (IDH-wildtype) and DIPG

  o DIPG patients must meet clinical and imaging requirements for DIPG diagnosis. Patients with newly diagnosed diffuse intrinsic pontine gliomas (DIPGs), defined as tumors with a pontine epicenter and diffuse involvement of 2/5 or more of the pons, are eligible without histologic confirmation. Patients with brainstem tumors that do not meet these criteria or not considered to be typical intrinsic pontine gliomas will only be eligible for Stratum B if the tumors have been biopsied and are proven to be an anaplastic astrocytoma, glioblastoma multiforme, gliosarcoma, anaplastic mixed glioma or fibrillary astrocytoma.
* Stratum 3: Low-grade glioma (IDH-wildtype) with multifocal/disseminated and/or leptomeningeal disease
* Stratum 4: Diffuse Leptomeningeal Glioneuronal Tumor
* Stratum 5: Pineoblastoma
* Stratum 6: All other eligible tumor types
* DISEASE STATUS: Participants will be eligible at any stage of disease.
* AGE: All children and adolescent/young adult (AYA) patients =< 21 years of age are eligible. AYA patients < 40 are eligible with a primary brain tumor entity more common in children than adults
* CEREBROSPINAL FLUID (CSF) COLLECTION: Patients must have a clinical indication for at least one CSF (lumbar, cisternal or ventricular) collection, or clinical circumstance where CSF sampling is feasible with no or minimal risk (e.g., endoscopic third ventriculostomy, external ventricular drain).
* INFORMED CONSENT: The patient or parent/guardian can understand the consent and is willing to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

* DIAGNOSIS: Given the extremely low rate of CSF cfDNA positivity in patients with localized, non-disseminated low-grade glioma, those patients will be excluded from participation.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will enroll from and be seen at Pediatric Brain Tumor Consortium sites and will meet the eligibility criteria in order to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2027-07-12 (Estimated); Study Completion 2028-07-12 (Estimated)

PRIMARY OUTCOMES:
Concordance of mutations across the tumor tissue vs. CSF | 3 months
  Within specific histologies with paired samples, estimate the concordance of mutation detected in the tumor tissue vs. cerebrospinal fluid cell free DNA (CSF cfDNA) across samples collected within 8 weeks of each other.

SECONDARY OUTCOMES:
Estimate the frequency of detection of CSF cfDNA across different types of pediatric CNS tumors in association with various disease states. | 3 months
  Intra-patient matched samples of CSF and tissue will be summarized for each oncogenic alteration and scored as positive vs. negative.
Track and estimate the correlation between the levels of CSF cfDNA and disease response as determined by clinical and imaging criteria across different disease types. | 3 months
  Associations between the quantity of cfDNA and standard clinical and imaging disease response will be assessed by either Wilcoxon rank-sum or Spearman's correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Miller, MD, PhD, Study Chair — NYU Langone Health
Locations (10):
- United States (9):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Lucille Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The Pediatric Brain Tumor Consortium (PBTC) ensures that high dimensional molecular data generated from PBTC samples will be submitted to the NIH Database of Genotypes and Phenotypes (dbGaP) or other NIH-designated data repository. PBTC is required to make data available to other investigators for use in research projects. An investigator requesting data from published PBTC studies will submit a proposal describing the studies from which data are requested, the requested data, and a list of investigators in the project and their affiliated institutions, along with the investigator's CV to the PBTC Steering Committee for review. Once approved, the requesting investigator will be asked to complete a Data Transfer Agreement before the release of deidentified data. Requests for data are typically only considered once the primary study manuscript has been published though exceptions may be made in the event of long delays in the primary study data publication.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after publication and end timeframe may be up to 10 years.